CLINICAL TRIAL: NCT02206919
Title: Magnetic Resonance Imaging of Vascular Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Dr. Alan Moody, Staff physician, Sunnybrook Health Sciences Centre
Other Study IDs: 066-2013
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes; Endothelial Dysfunction
Keywords: Flow mediated dilation; Magnetic Resonance Imaging MRI; Diabetes; Endothelial dysfunction; Popliteal artery; Atherosclerosis; Cardiovascular disease; Vascular disease
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A major function of blood vessels is to control blood flow by dilating or constricting depending on the demand. Vascular dysfunction is a state in which blood vessels fail to carry out its normal roles such as regulating blood flow. Diabetes is a risk factor for vascular dysfunction. Dysfunction may involve the smaller and/or larger blood vessels. Failure in the ability of large (conduit) blood vessels to control blood flow may be an early feature of atherosclerosis, a leading cause of stroke and heart attack. Measures of blood vessel dilation give an indication of the health of the vessel. Ultrasound and MRI can assess vascular function by measuring changes in blood vessel dilation. Diabetes may also affect tiny vessels in the kidney. These vessels become porous allowing albumin (a protein in the blood) to leak into the urine. The investigators can easily measure the presence of albumin in the urine.

This study aims to explore if MRI can demonstrate an association between vascular health in tiny and larger (conduit) blood vessels, by testing for an association between blood flow regulatory capacity of large vessels and presence of albumin in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with type 2 diabetes who:

  * are treated with oral hypoglycemic agents at a stable dose for at least 8 weeks
  * have diabetes diagnosed >6 months
  * have maintained stable weight for 2 months (within 3%)
  * have a valid Ontario Health Insurance Plan (OHIP) card and a family physician
  * if prescribed lipid medication, have taken a stable dose for at least 2 weeks
  * if prescribed blood pressure medication, have taken a stable dose for at least 1 week
  * can keep written food records
  * carotid intima-media thickness (cIMT) < 1.2 mm and ankle brachial index (ABI) of >0.9.

Exclusion Criteria:

* Individuals who

  * take insulin
  * take steroids
  * have GI disease (gastroparesis, celiac disease, ulcerative colitis, Crohn's Disease, IBS)
  * have had a major cardiovascular event (stroke or myocardial infarction) in the past 6 months
  * take warfarin (Coumadin)
  * have had major surgery in the past 6 months
  * have a major debilitating disorder
  * have clinically significant liver disease ( liver transaminase levels > 130 U/L), excluding Nonalcoholic fatty liver (NAFL) disease or NASH
  * have hepatitis B or C
  * have renal failure (high creatinine > 150 mmol/L)
  * have serum triglycerides ≥ 6.0 mmol/L
  * have a history of cancer, except non-melanoma skin cancer (basal cell, squamous cell)
  * have food allergies to study food components
  * have acute or chronic infections (bacterial or viral)
  * have chronic inflammatory diseases (e.g. rheumatoid arthritis, lupus; ulcerative colitis)
  * have other conditions which in the opinion of any of the investigators would make them unsuitable for the study
  * Any condition or circumstance which would prevent an individual from having an MRI (e.g. individuals with prostheses or metal implants, or those who are excessively claustrophobic)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Popliteal FMD MRI technique correlates with albuminuria in those with early diabetic disease | One year
  If this MRI technique is sensitive enough to demonstrate an association between flow mediated dilatation (FMD) of the popliteal artery and albuminuria, this will make a case for the use of the MRI technique in measuring effects of various interventions on vascular function.

SECONDARY OUTCOMES:
Blood measures related to cardiovascular disease and renal function | One year
Dietary risk factors related to chronic disease | One year

CONTACTS AND LOCATIONS:
Overall Officials: Alan Moody, DR, Principal Investigator — Sunnybrook Health Sciences Center; David Jenkins, DR, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada